CLINICAL TRIAL: NCT07030907
Title: A Phase 1a/b Study to Evaluate the Safety and Efficacy of OPB-101, an Autologous Mesothelin (MSLN) CAR T Cell Therapy With Antigen-dependent Expression of OUTSMART™ Designed IL-2 Cytokine in Platinum-resistant Ovarian Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of OPB-101 in Platinum-resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Outpace Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPB-101-OV-101A
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer Recurrent; Ovarian Cancer; Platinum Resistant Ovarian Cancer
Keywords: Outpace; Ovarian cancer; Advanced ovarian cancer; cell therapy; CAR T
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OPB-101 Treatment Arm (Experimental)
  Interventions: Biological: OPB-101

INTERVENTIONS:
Biological: OPB-101 — An autologous mesothelin (MSLN) CAR T cell therapy with antigen-dependent expression of OUTSMART designed IL-2 cytokine

SUMMARY:
The goal of this clinical trial is to learn if OPB-101 is safe in platinum resistant ovarian cancer participants and also to find the optimal dose of OPB-101.

Participants will have their own T cells modified in a laboratory and given back to them as OPB-101 in this one-time treatment. Participants will be in the hospital when they receive OPB-101 and then be checked at the clinical site frequently for the first few months.

DETAILED DESCRIPTION:
A phase 1a/b study to evaluate the safety and efficacy of OPB-101, an autologous mesothelin (MSLN) CAR T cell therapy with antigen-dependent expression of OUTSMART™ designed IL-2 cytokine in platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at the time of signing the informed consent form.
2. Histologically confirmed diagnosis of high grade serous epithelial ovarian, peritoneal, or fallopian tube cancer based on local histopathological findings.
3. Recurrent platinum-resistant disease defined as: Disease that has recurred within 6 months of the last receipt of platinum-based therapy.
4. Received at least 2 prior lines of systemic chemotherapy including a platinum-based chemotherapy.
5. Received prior therapy with a PARP inhibitor if the subject has a known germline or somatic BRCA1/2 mutation.
6. Measurable disease.
7. Consent to provide archived tumor tissue sample.
8. ECOG performance status of 0 or 1.
9. Adequate organ function.
10. Alkaline phosphatase ≤ 2.5 x ULN
11. ≤ Grade 1 dyspnea and oxygen saturation levels (SpO2) > 92% on room air.
12. LVEF ≥ 50%
13. Life expectancy of ≥ 3 months
14. Adequate venous access.
15. Negative screen for infectious disease markers.
16. Negative serum pregnancy test.
17. Abstain from heterosexual activity or to use 2 forms of effective methods of contraception.

Note: Other protocol defined inclusion criteria could apply

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breastfeeding.
2. Uncontrolled bacterial, fungal, or viral infections.
3. Active infection requiring systemic therapy.
4. Bleeding or thrombotic disorders or at risk for severe hemorrhage.
5. Any form of primary immunodeficiency.
6. Had an allogenic tissue/solid organ transplant.
7. Active autoimmune disease.
8. Concurrent treatment with systemic high dose corticosteroids.
9. Unresolved acute effects of any prior therapy.
10. Active invasive cancer other than the cancer under study.
11. Significant lung disease.
12. Clinically significant pericardial effusion.
13. Prior radiotherapy within 2 weeks of start of study intervention.
14. No major surgery within 28 days prior to enrollment.
15. Received investigational agents or tumor vaccines.
16. Received chemotherapy within the previous 3 weeks.
17. History of grade ≥ 3 ascites.
18. Active CNS involvement.
19. Received a live vaccine within 30 days prior to study treatment.
20. Received prior CAR T cell therapy.
21. Received prior mesothelin targeted therapy.
22. Dependent on intravenous hydration or total parenteral nutrition. Note: Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 30 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days
  Incidence of dose-limiting toxicities (DLTs)
Safety | 2 years
  Incidence of all treatment-emergent adverse events (TEAEs); Grade 3, 4, 5 TEAEs, serious adverse events (SAEs); deaths due to TEAEs and all deaths
Safety | 2 years
  To determine the maximum tolerated dose (MTD) of OPB-101 and/or recommended Phase 1b dose(s)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Roswell Park, Buffalo, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No